CLINICAL TRIAL: NCT02057263
Title: The Effect of Alendronate on the Immune Response to Hepatitis B Vaccine in Healthy Adults - a Randomized Placebo-controlled Pilot Study
Brief Title: The Effect of Alendronate on the Immune Response to Hepatitis B Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth L. Hohmann, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014-P-000040
Record Dates: First submitted 2014-02-04; First posted 2014-02-07 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis B
Keywords: Vaccine; Adjuvant; Bisphosphonates; Alendronate; Hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B | interventions — Alendronate; Diphosphonates; Hepatitis B Vaccines; Recombivax HB; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alendronate and Hepatitis B Vaccine (Experimental): Participants in the experimental arm will receive 4 alendronate doses during their Hepatitis B vaccination course.
  Interventions: Drug: Alendronate; Drug: Hepatitis B Vaccine
- Sugar Pill and Hepatitis B Vaccine (Experimental): Participants in the experimental arm will receive placebo doses during their Hepatitis B vaccination course.
  Interventions: Drug: Hepatitis B Vaccine; Drug: Placebo

INTERVENTIONS:
Drug: Alendronate — Participants will receive 4 doses of alendronate during the course of the study.
  Other Names: Fosamax; Bisphosphonate
  Arms: Alendronate and Hepatitis B Vaccine
Drug: Hepatitis B Vaccine — Participants will receive 3 Hepatitis B vaccinations, according to the schedule outlined by the CDC.
  Other Names: Recombivax
Drug: Placebo — Participants will receive 4 doses of placebo during the course of the study.
  Other Names: Sugar Pill
  Arms: Sugar Pill and Hepatitis B Vaccine

SUMMARY:
Vaccines are one of our most effective public health tools but many who need them don't respond well and are not protected. Adjuvants boost immune responses and are commonly included in vaccine preparations. Bisphosphonates are the most commonly prescribed treatment for osteoporosis and may represent a new class of adjuvant. Bisphosphonates are well tolerated with chronic administration and have very few adverse effects. Research suggests that these medications can stimulate the immune system.

Bisphosphonates are of special interest in populations with impaired immunity and an inability to amount protective antibody responses following immunizations. We propose a pilot study to evaluate the clinical relevance of this finding in humans. We will study the effect of bisphosphonates on quantitative humoral immune response to hepatitis B vaccine in healthy older volunteers who have not previously received this vaccine.

DETAILED DESCRIPTION:
Background: Immunization is one of the most beneficial and cost-effective disease prevention measures available, but is not always efficacious, especially in older and immunosuppressed populations. This commonly encountered failure to produce protective antibodies following immunization leaves large parts of the population vulnerable to serious morbidity and mortality resulting from potentially preventable communicable diseases. Bisphosphonates, a commonly prescribed treatment for osteoporosis that is well tolerated with few adverse effects, has recently been shown to enhance B cell expansion and antibody production after vaccination in mice, and may represent a new vaccine adjuvant.

Aims: The purpose of this project is to evaluate the effect of bisphosphonates on the immune response to vaccination in adults using two complementary research methodologies:

1. Evaluating the effect of bisphosphonates on quantitative humoral immune response to hepatitis B vaccine in healthy older volunteers through a randomized clinical trial.
2. Evaluating the effect of bisphosphonate treatment on protection against influenza and influenza-like illness after seasonal Influenza immunization in the adult population through a population-level retrospective analysis.

Methods: The first part of the study consists of a randomized, placebo-controlled pilot study in which 20 healthy adults 40-70 years of age who are seronegative for Hepatitis B, will be randomized to receive either two doses of intramuscular hepatitis B vaccine with alendronate or hepatitis B vaccine with placebo. The primary outcome evaluated will be quantitative anti-HB surface IgG antibody titers in the study group compared to the placebo group at week 8 and at 6 months. The second part of the study is a retrospective population based case-control study utilizing extensive available data repositories. Rates of influenza, influenza-like illness and lower respiratory tract infections per 1000 subjects will be ascertained and compared between study and control populations for each year, while adjusting for potential confounders.

ELIGIBILITY:
Inclusion Criteria:

* Subject willing to undergo hepatitis B vaccination AND be randomized to receive 4 doses of alendronate or placebo
* Age 40-70
* Able to consent for self - ascertained by physician assessment at time of history and exam.
* Chronic stable medical conditions, if well controlled on current therapies are allowed. For example individuals with well-controlled angina, hypertension, diabetes on oral agents, treated or past depression or anxiety, COPD, asthma, metabolic syndrome, NASH, mild chronic renal insufficiency, past history of malignancy, with no therapy for at least 5 years may be included.
* Willing to use contraception, if a woman of child-bearing potential (WOCBP)

Exclusion Criteria:

* Pregnant, breastfeeding or planning a pregnancy
* Prior Hepatitis B infection OR vaccination
* Autoimmune disorders of any kind (e.g. multiple sclerosis, rheumatoid arthritis, lupus, Psoriasis etc.)
* HIV or Hepatitis C seropositive
* Any known immunodeficiency (decompensated cirrhosis, HIV/AIDS, prior bone marrow transplant, or other known immunodeficiency)
* Patients on any immunosuppressive agents including systemic corticosteroids, calcineurin inhibitors, mTOR inhibitors, lymphocyte depleting biologic agents, anti-TNF agents, and others; chemotherapeutic anti-neoplastic agents within 5 years. Stable doses of inhaled corticosteroids for asthma/COPD are allowed.
* Gastroesophageal reflux disease (GERD), peptic ulcer disease, chronic proton pump inhibitors, chronic antacid use
* Chronic non-steroidal anti-inflammatory use; daily ASA for cardiac prophylaxis is allowed.
* Esophageal disorders of any kind
* Recent major dental work in the preceding 6 months, excluding dental cleaning and simple cavity filling
* History of jaw trauma
* Current or prior bisphosphonate use
* Prior history of severe reactions to vaccines
* Yeast or bisphosphonate allergy
* History of hypocalcemia
* Inability to stand or sit upright for at least 30 minutes.
* Any malabsorptive disorder including celiac disease, CF, Inflammatory bowel disease, recurrent C. difficile colitis, other colitis, prior gastrectomy, bariatric surgery or chronic diarrhea.
* Diabetes requiring insulin
* Body mass index > 31

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety/Adverse events | 5 months after final alendronate administration/second vaccination
  Safety is assessed by clinical symptoms and exam at final in-person visit. Standardized CTAE will be recorded and graded (mild/moderate/severe) with a special focus on vaccine related adverse events: Temperature, local injection site reactions, fatigue and malaise, AND adverse events related to alendronate which are primarily gastrointestinal: nausea, vomiting, esophagitis, ulceration. Rare, unlikely events such as atypical fractures and jaw osteonecrosis are extremely unlikely with this duration of dosing (4 weekly doses) but will also be specifically sought.

SECONDARY OUTCOMES:
Efficacy | 8 weeks to 5 months after final alendronate dose
  Efficacy is assessed by quantitative Anti Hepatitis B Surface IgG (immunoglobulin G) antibody titers in international units (iU) per ml. All subjects must have levels of ZERO in order to participate. A value of 10 iU/ml is considered protective. Titers directed against hepatitis B surface antigen will be measured by commercially available testing Efficacy will also be assessed as a categorical value: Yes/No for protective level of antibody achieved at either 8 weeks or 6 months (5 months after second vaccination). A protective level of hepatitis B surface antibody is defined as 10 iU/ml; levels of 10-100 are considered protective but "poorly responsive." We will compare mean titers between groups (placebo vs. alendronate). We believe a mean increase of 20% is likely clinically significant/important.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Available upon request